CLINICAL TRIAL: NCT06786260
Title: Di-PKD: A Pilot Trial of a 12-Month Targeted Dietary Intervention on Cyst Progression in Patients With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Di-PKD: A Pilot Trial of Dietary Intervention in Patients With Autosomal Dominant Polycystic Kidney Disease
Acronym: ADPKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5240615
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: ADPKD; Diet
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Diet (Experimental): Subjects will follow a specified diet (low salt, limited caffeine, high potassium, low phosphate, and limited protein and carbohydrate intake along with adequate water intake) after 1 week of preconditioning for 12 months.
  Interventions: Other: Interventional Diet
- Regular Diet (No Intervention): Subjects will follow the diet they normally adhere to after 1 week of preconditioning.

INTERVENTIONS:
Other: Interventional Diet — Low salt, limited caffeine, high potassium, low phosphate, and limited protein and carbohydrate intake along with adequate water intake diet
  Arms: Interventional Diet

SUMMARY:
The goal of this interventional study is to evaluate the impact of a specific diet (low salt, limited caffeine, high potassium, low phosphate, limited protein, limited carbohydrate intake, adequate water intake) on changes in serum and urinary biomarkers, total kidney volume (TKV), and cyst progression in subjects with autosomal dominant polycystic kidney disease (ADPKD).

Researchers will compare the results of subjects in the study diet (interventional) arm to the results of subjects in the regular diet (control) arm.

DETAILED DESCRIPTION:
15 subjects will be enrolled in each dietary arm for a total of 30 subjects. All subjects will follow the study diet for one week, after which serum and urinary biomarkers will be measured. A baseline evaluation, including genetic testing, MRI, Mayo Clinic Imaging Classification and 10-question survey will also be conducted. After Week 1 of the study, subjects will be assigned to the intervention or control arm. Subjects will have six follow-up visits at months 1, 2, 3, 6, 9 and 12 to assess adherence to diet. Serum and urinary biomarkers will be repeated at each visit. MRI will be repeated at Month 12.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ADPKD
* Genetic testing confirmation of PKD1 or PKD2
* eGFR >30mL/1.73m2
* Willingness to adhere to a preconditioning diet for 1 week and ability to complete the study
* Mayo Clinic Imaging Classification (MCIC): 1C, 1D, 1E

Exclusion Criteria:

* History of dietary non-adherence
* Subjects on Tolvaptan
* Comorbidities that could interfere with participation (Diabetes, Heart Failure (EF<30%) Advanced Chronic Kidney Disease (CKD) Stage 4 and higher)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Progression of kidney cysts by change in total kidney volume (TKV) from baseline to 12 months | Change between baseline and 12 months
  A composite measurement of MRI to determine total kidney volume (TKV) by kidney length, width, and depth will be done at baseline and again at 12 months. MRI results will be compared between the two-time points to assess the cyst progression, if any. An increase of about 5% per year from baseline will be significant.

SECONDARY OUTCOMES:
Progression of kidney cysts as evidenced by urinary biomarkers from baseline to 12 months | Change between baseline and 12 months
  A urine sample will be collected at the end of the preconditioning week to establish a baseline for the urinary biomarkers cAMP and MCP-1. This is a composite measurement. Values for cAMP and MCP-1 at 12 months will be compared to the baseline values. If the values at 12 months remain the same or less than the composite baseline values, this will indicate a low likelihood that the kidney cysts have progressed. A significant change of 20% or greater overall in the combined biomarkers will indicate a kidney cyst progression.
Progression of kidney cysts as evidenced by serum biomarkers from baseline to 12 months | Change between baseline and 12 months
  A blood draw will be performed at the end of the preconditioning week to establish a baseline for the serum biomarkers uric acid, ADH, FGF-23, bicarbonate, and cystatin C. This is a composite measurement. Values for uric acid, ADH, FGF-23, bicarbonate, and cystatin C at 12 months will be compared to the baseline values. If the values at 12 months remain the same or less than the composite baseline values, this will indicate a low likelihood that the kidney cysts have progressed. A significant change of 20% or greater overall in the combined biomarkers will indicate a kidney cyst progression.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Abdipour, MD, Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No